CLINICAL TRIAL: NCT04221334
Title: Clinical Investigation Examining Plaque and Gingivitis Reductions of Connected Toothbrush Compared to Non-Connected Toothbrush: a Six-week Clinical Study in California
Brief Title: Clinical Investigation Examining Plaque and Gingivitis Connected Toothbrush Compared to Non-Connected Toothbrush
Acronym: Connected
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRO-2018-12-CTB-PLA-LLU-YPZ
Record Dates: First submitted 2019-09-30; First posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Gingivitis; Plaque, Dental
MeSH Terms: conditions — Gingivitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Product Code: XX Brush twice daily (morning and evening) for at least 2 minutes each time Cover the entire length of bristles with toothpaste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental Toothbrush 1 (Active Comparator): 1. A connected power toothbrush; brushed twice daily (morning and evening) for two (2) minutes, with Colgate Cavity Protection Toothpaste; Oral.
  Interventions: Device: Electric Toothbrush; Other: oral health care application
- Experimental Toothbrush 2 (Active Comparator): 2. A non-connected power toothbrush; brushed twice daily (morning and evening) for two (2) minutes, with Colgate Cavity Protection Toothpaste; Oral.
  Interventions: Device: Electric Toothbrush

INTERVENTIONS:
Device: Electric Toothbrush — Electric Toothbrush used to remove dental plaque and resolve gingivitis
Other: oral health care application — phone application that shows the user brushing efficiency real time
  Arms: Experimental Toothbrush 1

SUMMARY:
The objective of this clinical research study is to assess plaque and gingivitis reductions of Connected Toothbrush compared to Non-Connected Toothbrush over a six-week clinical study.

DETAILED DESCRIPTION:
A phase II randomized, single-center, two-cell, examiner-blind and parallel-group clinical study conducted in the Loma Linda, California area, to investigate the clinical efficacy of a connected power toothbrush as compared to a non-connected power toothbrush in reducing dental plaque and gingivitis as measured by the Rustogi Modification of the Navy Plaque Index and Löe and Silness Gingival Index over a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

1. • Male and female subjects had to be between the ages of 18 and 70 (inclusive),
2. • Subjects needed to be available for the duration (6 weeks) of the study,
3. • Subjects had to possess minimum of 20 uncrowned permanent natural teeth (excluding third molars),
4. • Subjects were required to present and an initial mean gingivitis score of at least 1.0 as determined by the use of the Löe-Silness Gingival Index,
5. • Subjects were required to present an initial mean plaque index of at least 0.6 as determined by the use of the Rustogi Modification of the Navy Plaque Index,
6. • Subjects had to sign an Informed Consent form,
7. • Subjects had to be in general good health and
8. • Subjects with no known history of allergies to personal care/consumer products or their ingredients, relevant to any ingredients in the test products as determined by the dental/medical professional monitoring of the study.

Exclusion:

1. • Medical condition which require pre-medication prior to dental visits/procedures,
2. • The presence of partial removable dentures,
3. • Subjects who had advanced periodontal disease (gum disease),
4. • Five (5) or more decayed or untreated dental sites at screening (cavities),
5. • Subjects with diseases of the soft or hard oral tissues,
6. • Subjects with orthodontic appliances/bands/lingual bars that interfere with any clinical assessment (plaque scoring),
7. • Dry mouth as a result of a medication or medical condition,
8. • Use of drugs that can currently affect salivary flow,
9. • Use of antibiotics one (1) month prior to or during this study,
10. • Use of any over the counter medications other than analgesics that could interfere with the study at PI discretion,
11. • Chronic (>3 3 times/week) use of medications that are known to affect gingival tissues including steroids or non-steroidal anti-inflammatory medications or the listed medications (phenytoin, calcium antagonists, Coumadin, cyclosporine),
12. • Any diseases that might affect the assessment of the study treatment or gingival tissues (rheumatoid arthritis, Crohn's disease, diabetes), ongoing chemotherapy for cancer, radiation therapy for head and neck cancer,
13. • Pregnant or breast-feeding women were excluded from the study,
14. • Subjects who participated in any other clinical study in the month preceding this study,
15. • Allergic to common dentifrice ingredients,
16. • Medical condition which prohibits not eating/drinking or chewing gum for 4 hours prior to their scheduled visit,
17. • Immune compromised individuals (AIDS, immune suppressive drug therapy) and
18. • History of infectious disease or other blood borne diseases (Hepatitis series, HIV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
change in mean dental plaque | 3 and 6 weeks of product use
  Reduction in plaque measurement is served as primary efficacy variable toothbrush for 6 weeks for each subject.
change in mean gingivitis | 3 and 6 weeks of product use
  gingivitis measurement is served as secondary efficacy variable

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Yi, DDS/PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No